CLINICAL TRIAL: NCT03438201
Title: The Efficiency of Different Amount of Protein Intake Associated With a Physical Activity Protocol in Surgical Cancer Patients Admitted to the Intensive Care Unit : Randomized Controlled Trial
Brief Title: Protein Intake Associated With Physical Activity Related to Specific Outcomes
Acronym: STRENGTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliano P Almeida, MD, PhD, Medical Doctor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77623917.0.0000.0065
Record Dates: First submitted 2018-01-29; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cancer; Critically Ill; Surgery
Keywords: Cancer, ICU, Surgery, Protein, Physical Activity
MeSH Terms: conditions — Neoplasms; Critical Illness; Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-protein diet (Active Comparator): High Protein Diet (2,0 - 2,5g/Kg body weight/day) Physical Activity protocol
  Interventions: Dietary Supplement: Intervention
- Normoproteic diet (Active Comparator): Standard Protein Diet (1,0 - 1,2g/Kg body weight/day) Physical Activity protocol
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Intervention — Enteral feeding that will give the patient the amount of protein between 2.0 - 2.5 Kg/body weight/Day
  Other Names: High Protein intake
  Arms: High-protein diet
Dietary Supplement: Control — Enteral feeding that will give the patient the amount of protein between 1.0 - 1.2 Kg/body weight/Day
  Other Names: Standard Protein Intake
  Arms: Normoproteic diet

SUMMARY:
This is a Randomized Controlled Trial . The purpose of this study is to assess the hypothesis that whether a high protein diet combined with a physical activity protocol in surgical cancer patients admitted to the ICU in the post operative period is associated with better physical function at the hospital discharge as well as a better quality of life.

DETAILED DESCRIPTION:
Surgical cancer patients will be categorized by their nutritional risk using a specific screening toll. During the hospital stay some measurements will be done. Such as resting energy expenditure (REE) before and after surgery; physical function evaluation; strength and quality of life.

The proposed intervention is a post operative diet with a different amount of protein (diet with a standard amount of protein and a diet with high amount of protein) associated to an institutional protocol of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Age greater than or equal to 18 years old
* Have a tendency to be admitted to the ICU after the surgery
* Fill the eligible criteria to start enteral feeding within 72 hours
* Sign the consent form;

Exclusion Criteria:

* Mechanical ventilation such as fraction of inspired oxygen inspired oxygen fraction (FiO2) >60% or positive end expiratory pressure (PEEP) > 12cm H2O
* Bronchopleural fistula
* Karnofsky <50
* Participant cannot b enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-04-04 (Estimated); Primary Completion 2018-10-12 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Physical Function | 8 days after randomization
  6 minutes walk test

SECONDARY OUTCOMES:
Physical Function | 30 days after randomization
  6-minute walk test after 30 days the date of randomization;
Quality of life | 6 months after randomization
  Measurement of quality of life using the Euro-Qol 5D-5L index. EQ-5D-5L index includes five questions concerning mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A summary utility index value can be computed from subject's response to these five questions. Values range from -0.594 (worst possible health score) to 0 (death) to 1.000 (best health).
Body Composition related to prognosis | 8 days after randomization
  Phase Angle (BIA)
Postoperative complications | 30 days after randomization
  Clavien Dindo
Resting Energy Expenditure | one day before surgery and one day after surgery
  Indirect Calorimetry
Length of hospital stay. | 30 days after randomization
  Starts in the first day of hospitalization and ends on the day of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Juliano P Almeida, Professor, Principal Investigator — University of Sao Paulo; Ilana Roitman, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculty of Medicine University of Sao Paulo, São Paulo, São Paulo, Brazil